Study protocol & Statistical analyses plan

Official title: Digitally Supported Intervention to Master Complex Fall Risk

Situations in Persons with Multiple Sclerosis – a Multicenter Study (STAR)

Brief title: Intervention to Master Complex Fall Risk Situations in Persons

with Multiple Sclerosis (STAR)

Protocol date: 2025-12-0812-08 ID 285079

**Background** Fifty-six percent of those with a mild to moderate multiple sclerosis (MS) report

falls during a three-month period and 60 % express fear of falling. Several fall risk factors have

been identified a complexity of falls including the interaction of triggering factors and

preceding activities and events has been described. There is a lack of studies explicitly

evaluating fall prevention strategies given as counselling over time.

Methods This is a two-armed internal pilot study with a parallel group design and random

allocation to control or intervention group (1:1). The pilot study will evaluate feasibility in

terms of recruitment, drop-outs, adverse events and battery of tests, and constitute the base for

recalculation of the beforehand estimated sample size for a full-scale study. The full-scale study

will evaluate whether a fall preventative strategy based on individual fall risk evaluation will

reduce fall frequency compared to general fall preventative information. The hypothesis is that

the intervention group will report 30% less falls during the 6-months period when the

intervention is active, compared to the control group. Based on descriptions of recent fall

situations, fall risk factors will be categorized using the International Classification of

Functioning, Disability and Health. Participants in the intervention group will discuss the

impact from specific MS-symptoms, environmental and personal factors, triggering factors and

activities and/ or circumstances that the individual perceive precede fall situations with the

physiotherapist leading to individual strategies. The control group will receive general fall risk

prevention recommendations. After completion of the study, the control group will be offered individual strategies based on reported falls.

Adults diagnosed with MS, fall history and remained walking ability will be recruited in six sites in Sweden by physiotherapists. Primary outcome is self-reported falls during six months. Secondary outcomes are self-rating scales focusing on concern of falling, confidence in remaining balance during activities, walking limitations and ability to avoid falls.

able 1. Participant timeline: Schedule of enrollment, interventions, and assessments.

| | TRIAL PERIOD | | | |
|---|---|---|---|---|
| | Enrollment | Allocation | Post-randomization | Follow-up |
| IIMEPOINT | - <u>t</u> , | <b>t</b> ∂ | t <sub>2</sub><br>For 6 months | tı |
| ENROLLMENT: | | | | |
| Eligibility screen | Х | | | |
| Informed consent | Х | | | |
| Check for inclusion and exclusion<br>criteria | | Х | | |
| Randomization | | Х | | |
| INTERVENTION/ COMPARATOR: | | | | |
| Individual fall preventative strategy<br>as add-on to general fall risk<br>information] | | Х | | |
| General fall risk information | | Х | | |
| ASSESSMENTS: | | | | |
| Demographic data *, Timed Up and<br>Go test, Six Spot Step test, Symbol<br>Digit Modalities test, 29-item MS<br>Impact scale | | Х | | |
| Number of falls, falls description,<br>injury due to fall, need to seek care | | , | | |
| due to fall, adverse events. | | Х | Every two weeks. | |
| Falls Efficacy scale International, Activities-specific Balance Confidence scale, 12-item MS Walking scale, Frändin Grimby Physical activity scale, Fear of falling, Avoid activities due to fall risk, Master fall risk, Understanding fall risk factors, Self-rated change in balance | | х | | х |

<sup>\*</sup>Sex, gender, MS-type, falls last 3 months, ongoing physiotherapy/rehabilitation, walking device, occupation, living condition, contact information\*\*exacerbation, ongoing physiotherapy/rehabilitation, changes in walking device use, living condition or occupation

## Statistical methods

The flow of participants through the study will be examined and illustrated according to the Consolidation Standard of Reporting Trials (CONSORT) (1). We will calculate the proportion of participants lost to follow-up.

Analyses will be performed on an intention-to-treat basis. Baseline demographic and clinical characteristics of the study participants will be summarized for the two intervention groups separately. Continuous variables will be summarized using the measures of central tendency and dispersion (mean and standard deviation, the median and interquartile range as well as minimum and maximum values) as appropriate based on the distribution. Categorical variables will be summarized using frequencies and percentages. Since baseline characteristics are expected to be balanced between intervention groups due to randomization, we will evaluate if any substantial imbalance may have occurred by chance.

The distribution of outcome data will be examined. For the analysis of primary outcome, we will consider Poisson regression if the assumptions are satisfied or Negative binomial regression, which relaxes the assumption made by Poisson regression that the variance is equal to the mean. We may consider also Cox regression to compare time to the first fall between intervention arms. Since falls may occur repeatedly in patients with MS, we may consider also extensions of Cox proportional hazards regression that are for recurrent event analyses. Estimates unadjusted and adjusted for baseline covariates will be presented. Secondary outcomes will be analyzed according to the measurement type and distribution.